CLINICAL TRIAL: NCT04740047
Title: Cios Mobile 3D Spin for Robotic Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Intuitive Surgical (Industry); Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Principal Investigator, Janani S. Reisenauer, Principal Investigator, Mayo Clinic
Other Study IDs: 20-004757
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Nodule, Solitary; Pulmonary Cancer; Lung Cancer; Lung Cancer, Nonsmall Cell; Lung Adenocarcinoma
MeSH Terms: conditions — Solitary Pulmonary Nodule; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pulmonary Nodule: Pulmonary nodule is suitable for elective bronchoscopy with a moderate to high risk of lung cancer based on clinical, demographic and radiologic information or with suspected metastatic disease.
  Interventions: Diagnostic Test: Ion Endoluminal System

INTERVENTIONS:
Diagnostic Test: Ion Endoluminal System — Robotic bronchoscopy with c-arm imaging.
  Other Names: Cios 3D mobile spin system

SUMMARY:
Evaluate the clinical utility and early performance of the Cios 3D Mobile Spin in conjunction with the Ion Endoluminal System, to visualize and facilitate the sampling of pulmonary nodules between 1-3 cm via the airway.

ELIGIBILITY:
Inclusion Criteria:

* Subject age 18 years and older
* Subject is suitable for elective bronchoscopy
* Subject with a moderate to high risk of lung cancer based on clinical, demographic and radiologic information or with suspected metastatic disease
* Solid or semi-solid pulmonary nodules of ≥ 1cm and ≤3.5 cm in largest dimension
* Nodule is located in bronchial generation 4+ (i.e. beyond segmental bronchus)
* Subject is a candidate for CT-guided needle biopsy
* Subject is able to understand and adhere to study requirements
* Subject is able to understand and adhere to study requirements and able to provide informed consent
* Subject is not legally incapacitated or in legal/court ordered institution
* Subject has no dependency on the investigator or sponsor

Exclusion Criteria:

* Lack of fitness or exercise capacity to undergo bronchoscopy under general anesthesia as determined by physician prior to procedure
* Acute myocardial infarction or unstable angina ≤ 6 weeks prior to study procedure
* Clinically relevant partial trachea obstruction or obstruction of vena cava per physician assessment
* Acute respiratory failure, clinically significant hypoxemia, or high respiratory rate (i.e. > 30 breaths per minute) per physician assessment
* Renal insufficiency that presents risk per physician's discretion or liver failure (i.e. CHILD-PUGH Class C)
* World Health Organization functional Class IV Pulmonary Hypertension or history of clinically significant mPAP
* Known or suspected pregnancy
* Recent head injury (<12 weeks pre-procedure) or subjects presenting with clinically significant neurologic deficits
* Unstable hemodynamic status (i.e. Dysrhythmia requiring intervention, altered mental status/consciousness)
* Inability to adequately oxygenate subject during procedure per physicians discretion (i.e. unable to achieve S02 > 88% or requiring >4L of oxygen prior to procedure)
* Subject with uncorrectable coagulopathy, bleeding or platelet disorders, history of major bleeding with bronchoscopy
* Subjects contraindicated for intubation or general anesthesia, or subjects with ASA ≥ 5
* Subjects taking antiplatelet (i.e. clopidogrel), anti-coagulant (i.e. heparin or warfarin) or /platelet aggression inhibitors (i.e. Abciximac or Eptifibatide) medications that cannot be stopped per standard practice, i.e. 5-7 days pre-procedure or heparin that cannot be held according to standard practice (6-12 hours). Aspirin not included.
* Any severe or life-threatening comorbidity that could increase the risk of bronchoscopic biopsy
* Moderate-to-severe pulmonary fibrosis presenting procedural risk as assessed by physician
* Endobronchial lesion associated with lobar atelectasis
* Known allergy, sensitivity or previous allergic reaction to ortho-phthalaldehyde (OPA)
* Non-systemic treatment for lung cancer (i.e. SBRT) performed in the same lobe as the target nodule(s)
* Previous surgical intervention performed in the same lobe as the target nodule (s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from pulmonary, medical oncology or thoracic surgery departments at the Mayo Clinic Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Tool in Lesion | At the time of the procedure
  Ability to visualize on 3D imaging the pre-planned target location characterized when displayed distance of catheter tip to nearest edge of the virtual target is ≤ 2cm and is oriented towards the lesion in 3 axes.

SECONDARY OUTCOMES:
Procedure-related complications | 6 months
  Overall incidence of procedure-related complications recorded as adverse events.
Duration-related outcomes | At the time of the procedure
  Reporting of times related to procedure times including procedure time, navigation time, time to 3D confirmation, time to tissue acquisitions, anesthesia time, and fluoroscopy time and dose.

CONTACTS AND LOCATIONS:
Overall Officials: Janani Reisenauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reisenauer J, Duke JD, Kern R, Fernandez-Bussy S, Edell E. Combining Shape-Sensing Robotic Bronchoscopy With Mobile Three-Dimensional Imaging to Verify Tool-in-Lesion and Overcome Divergence: A Pilot Study. Mayo Clin Proc Innov Qual Outcomes. 2022 Apr 23;6(3):177-185. doi: 10.1016/j.mayocpiqo.2022.02.004. eCollection 2022 Jun. PMID 35509435